CLINICAL TRIAL: NCT03497585
Title: Developing an Activity Pacing Framework for the Management of Chronic Pain/Fatigue. Stage III: Feasibility and Acceptability Studies
Brief Title: Developing an Activity Pacing Framework: Feasibility and Acceptability
Status: Completed | Type: Observational
Sponsor: Pennine Acute Hospitals NHS Trust (Other)
Collaborators: University of Leeds (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Deborah Antcliff, Senior Physiotherapist/Researcher, Pennine Acute Hospitals NHS Trust
Other Study IDs: IRAS:242203, V2.1, 27.04.18
Record Dates: First submitted 2018-03-23; First posted 2018-04-13 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain; Fibromyalgia; Chronic Fatigue Syndrome; Chronic Low Back Pain
Keywords: Rehabilitation; Pain Management
MeSH Terms: conditions — Chronic Pain; Fibromyalgia; Fatigue Syndrome, Chronic; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Activity Pacing Framework: Adult patients attending rehabilitation programmes underpinned by the activity pacing framework.
  Interventions: Behavioral: Activity pacing framework

INTERVENTIONS:
Behavioral: Activity pacing framework — The activity pacing framework will be used to structure and standardise the instructions of pacing in existing rehabilitation programmes for adult patients with chronic pain/fatigue. The activity pacing framework has been developed in Stages I and II of this research. Stage I involved an online survey of activity pacing across healthcare professionals in England. The survey findings, together with existing research were used to develop the first draft of the framework. The framework was refined in Stage II: Nominal group technique (consensus method). The activity pacing framework describes the aims, facets and stages of pacing, together with how pacing relates to different behavioural typologies and other pain management strategies.

SUMMARY:
This study explores whether it is feasible to use a newly developed activity pacing framework to standardise how activity pacing is instructed by healthcare professionals in rehabilitation programmes for patients with chronic pain/fatigue.

DETAILED DESCRIPTION:
Activity pacing is frequently advised in the management of chronic pain/fatigue, including chronic low back pain, chronic widespread pain/fibromyalgia and chronic fatigue syndrome/myalgic encephalomyelitis. However, there is no agreed definition of 'activity pacing' and it is instructed in various ways. For some, pacing involves adapting/limiting activities (for example, breaking down tasks/having rests); while for others, pacing involves having consistent activities/gradually increasing activities. Furthermore, pacing has been associated with both improved symptoms (decreased fatigue/anxiety/depression) and worsened symptoms (increased pain/disability).

Due to the high prevalence and cost (personal and financial) of chronic pain/fatigue, it is imperative that coping strategies such as pacing are clearly defined and evidence-based. This study involves Stage III in the development of an activity pacing framework to standardise how pacing is instructed by healthcare professionals. Stage I: Online Survey of pacing involved 92 healthcare professionals (doctors/nurses/physiotherapists/occupational therapists/clinical psychologists). The survey findings, together with existing research were used to develop the pacing framework. The framework was further developed in Stage II: Nominal Group Technique (consensus meeting), involving four patients and six healthcare professionals.

Stage III will test the feasibility of implementing the pacing framework clinically, by using it to underpin existing rehabilitation programmes for chronic pain/fatigue. Patients will attend rehabilitation programmes at the study sites as per usual practice. Patients' participation in this study involves their completion of a booklet of questionnaires. The aim of this feasibility study is to explore whether the activity pacing framework is usable in the clinical setting, to explore recruitment/retention rates, together with changes in symptoms between the start and end of treatment, and at 3-months follow-up. Stage III will also explore the acceptability of the framework by undertaking interviews with the patients and healthcare professionals involved in the rehabilitation programmes. Stage III is expected to last 22 months.

Future study will test the framework in a clinical trial to assess the effects of pacing on patients' symptoms. The pacing framework has the potential to improve treatments by providing guidance on the components of pacing found to have benefits for patients.

This study is funded by a Health Education England/National Institute for Health Research (HEE/NIHR) Integrated Clinical Academic (ICA) Clinical Lectureship.

ELIGIBILITY:
Feasibility Study Inclusion Criteria:

* Patients with an initial General Practitioner (GP)/hospital consultant referral to The Pennine Acute Hospitals NHS Trust with diagnoses of chronic low back pain, chronic widespread pain, fibromyalgia or CFS/ME, with a minimum symptom duration of 3 months.
* Patients referred to a rehabilitation programme for chronic pain/fatigue
* Patients aged ≥18 years
* Patients able to read/write in English

Exclusion Criteria:

* Patients with evidence of a serious underlying pathology, such as a current diagnosis of cancer
* Patients with severe mental health/cognitive functioning issues

Acceptability Study (qualitative interviews) Inclusion Criteria:

* Patients with an initial GP/hospital consultant referral to The Pennine Acute Hospitals National Health Service (NHS) Trust with diagnoses of chronic low back pain, chronic widespread pain, fibromyalgia or CFS/ME, with a minimum symptom duration of 3 months (as per the feasibility study).
* Patients who attended a minimum of one session of the rehabilitation programme, who consented to the study and completed the first questionnaire booklet. Patients do not need to have completed the programme, since the interviews will include patients who both completed and did not complete the programme.
* Qualified healthcare professionals delivering the rehabilitation programmes who received training in using the activity pacing framework: physiotherapists and psychological wellbeing practitioners employed by The Pennine Acute Hospitals NHS Trust and Pennine Care NHS Foundation Trust.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population involves patients with conditions of chronic pain/fatigue, for example, chronic low back pain, chronic widespread pain, fibromyalgia and chronic fatigue syndrome/myalgic encephalomyelitis (CFS/ME). The study population includes those patients who are referred to the physiotherapy departments of The Pennine Acute Hospitals National Health Service (NHS) Trust and who attend a rehabilitation programme. The activity pacing framework will be used to structure and standardise the pacing component of the programme.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Antcliff, PhD, BSc, Principal Investigator — Pennine Acute Hospitals NHS Trust
Locations (1):
- The Pennine Acute Hospitals NHS Trust, Bury, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Antcliff D, Campbell M, Woby S, Keeley P. Activity Pacing is Associated With Better and Worse Symptoms for Patients With Long-term Conditions. Clin J Pain. 2017 Mar;33(3):205-214. doi: 10.1097/AJP.0000000000000401. PMID 27322396
- [Derived] Antcliff D, Keenan AM, Keeley P, Woby S, McGowan L. Testing a newly developed activity pacing framework for chronic pain/fatigue: a feasibility study. BMJ Open. 2021 Dec 8;11(12):e045398. doi: 10.1136/bmjopen-2020-045398. PMID 34880007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the feasibility study, patient recruitment occurred between 21st May 2018 and 3rd September 2019. Patients were recruited from those referred to a rehabilitation programme within a physiotherapy-led, out-patient service in a National Health Service (NHS) Trust in Northern England.
  The acceptability interviews involved patients (as above) and healthcare professionals (HCPs) delivering the programmes. HCP recruitment occurred between 18th September 2019 and 6th November 2019.
Pre-assignment Details: This was a single-arm feasibility study. All patients received the same treatment, that is, they all attended the same rehabilitation programme that was underpinned by the activity pacing framework. Excluded from the study were those patients who did not meet the inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Activity Pacing Framework
Started | 112 (112 participants were recruited: 107 patients, plus 5 HCPs for the acceptability interviews.)
Completed | 57
Not Completed | 55

BASELINE CHARACTERISTICS:
Population: All 107 participants were included in the baseline analyses. Some questions have fewer than 107 responses in instances of missing answers. For the question regarding participants' conditions, they were able to check more than one answer.
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One missing answer
  years
    number analyzed (Participants) | 106
    (all) | 55.25 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One missing answer
  Participants
    Ethnicity: number analyzed (Participants) | 106
    Ethnicity: White (British, Irish, Other) | 99
    Ethnicity: Black (Caribbean, African) | 1
    Ethnicity: Mixed (White/Black, White/Asian, other) | 3
    Ethnicity: Asian (Indian, Pakistani, Bangladeshi, other) | 3
    Ethnicity: Asian Eastern (Chinese, other) | 0
Conditions [Count of Participants; unit: Participants] — Participants could check more than one condition in the tick box. Population: One participant gave a missing answer
  Participants
    Low back pain: number analyzed (Participants) | 106
    Low back pain | 79
    Chronic widespread pain: number analyzed (Participants) | 106
    Chronic widespread pain | 52
    Fibromyalgia: number analyzed (Participants) | 106
    Fibromyalgia | 29
    Chronic fatigue syndrome/myalgic encephalomyelitis (CFS/ME): number analyzed (Participants) | 106
    Chronic fatigue syndrome/myalgic encephalomyelitis (CFS/ME) | 12
    Other (e.g. osteoarthritis): number analyzed (Participants) | 106
    Other (e.g. osteoarthritis) | 21
Number of conditions [Count of Participants; unit: Participants] — Number of the above conditions (multiple co-morbidities) Population: One missing answer
  Participants
    number analyzed (Participants) | 106
    1 condition | 41
    2 conditions | 49
    3 conditions | 12
    4 conditions | 2
    5 conditions | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Activity Pacing Questionnaire (APQ-28) From Baseline to the End of the 6-week's Programme
Description: The Activity Pacing Questionnaire (APQ) was developed to measure different themes of activity pacing. The APQ was initially validated among a sample of patients with chronic pain/fatigue and contained 26 items. Factor analysis identified five themes of pacing contained within the APQ-26: Activity adjustment, Activity consistency, Activity planning, Activity acceptance and Activity progression.
  The APQ-26 has been modified for the purpose of this study with the addition of two items to correspond to important aspects of pacing that were not included in the APQ-26. The APQ-28 reflects the content of the activity pacing framework.
  The APQ-28 will be used to assess the changes in activity pacing from baseline (pre-treatment: up to one week before the programme) to end of the programme (6-week's programme).
  Each of the five themes of pacing is calculated as a mean score (0-4), where higher scores indicated more implementation of pacing strategies.
Time Frame: Change in activity pacing from baseline (pre-treatment: up to one week before the programme) to the end of the 6-week's programme
Population: Of the 107 participants who commenced the rehabilitation programme and provided baseline data (T1), 65 participants completed the data collection at the end of the 6-week rehabilitation programme. There were two missing answers for APQ-28 Activity adjustment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 65
score on a scale
  APQ-28 Activity adjustment: number analyzed (Participants) | 63
  APQ-28 Activity adjustment | 0.70 [0.48 to 0.91]
  APQ-28 Activity planning | 0.99 [0.72 to 1.26]
  APQ-28 Activity consistency | 0.84 [0.60 to 1.07]
  APQ-28 Activity acceptance | 0.67 [0.46 to 0.89]
  APQ-28 Activity progression | 0.94 [0.65 to 1.22]

2. Secondary Outcome: Activity Pacing at Baseline: Activity Pacing Questionnaire (APQ-28)
Description: The Activity Pacing Questionnaire (APQ) was developed to measure different themes of activity pacing. The APQ was initially validated among a sample of patients with chronic pain/fatigue and contained 26 items. Factor analysis identified five themes of pacing contained within the APQ-26: Activity adjustment, Activity consistency, Activity planning, Activity acceptance and Activity progression.
  The APQ-26 has been modified for the purpose of this study with the addition of two items to correspond to important aspects of pacing that were not included in the APQ-26. The APQ-28 reflects the content of the activity pacing framework.
  The APQ-28 will be used to measure activity pacing at baseline (pre-treatment: up to one week before the programme).
  Each of the five themes of pacing is calculated as a mean score (0-4), where higher scores indicated more implementation of pacing strategies.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: Included in these analyses are all 107 participants who provided data at baseline. There is one missing answer for APQ-28 Activity adjustment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 107
score on a scale
  APQ-28 Activity adjustment: number analyzed (Participants) | 106
  APQ-28 Activity adjustment | 1.83 (0.81)
  APQ-28 Activity planning | 1.49 (0.98)
  APQ-28 Activity consistency | 1.85 (0.94)
  APQ-28 Activity acceptance | 1.91 (0.92)
  APQ-28 Activity progression | 1.51 (0.95)

3. Secondary Outcome: Activity Pacing at the End of Treatment: Activity Pacing Questionnaire (APQ-28)
Description: The Activity Pacing Questionnaire (APQ) was developed to measure different themes of activity pacing. The APQ was initially validated among a sample of patients with chronic pain/fatigue and contained 26 items. Factor analysis identified five themes of pacing contained within the APQ-26: Activity adjustment, Activity consistency, Activity planning, Activity acceptance and Activity progression.
  The APQ-26 has been modified for the purpose of this study with the addition of two items to correspond to important aspects of pacing that were not included in the APQ-26. The APQ-28 reflects the content of the activity pacing framework.
  The APQ-28 will be used to measure activity pacing at the end of the 6-week's programme.
  Each of the five themes of pacing is calculated as a mean score (0-4), where higher scores indicated more implementation of pacing strategies.
Time Frame: 6-weeks (end of the programme)
Population: Of the 107 participants who completed baseline data (T1), 65 completed data collection at the end of the 6-week rehabilitation programme (T2). There were two missing answers for APQ-28 Activity adjustment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 65
score on a scale
  APQ-28 Activity adjustment: number analyzed (Participants) | 63
  APQ-28 Activity adjustment | 2.43 (0.73)
  APQ-28 Activity planning | 2.42 (0.87)
  APQ-28 Activity consistency | 2.65 (0.74)
  APQ-28 Activity acceptance | 2.55 (0.72)
  APQ-28 Activity progression | 2.39 (0.89)

4. Secondary Outcome: Activity Pacing at 3-months Follow up: Activity Pacing Questionnaire (APQ-28)
Description: The Activity Pacing Questionnaire (APQ) was developed to measure different themes of activity pacing. The APQ was initially validated among a sample of patients with chronic pain/fatigue and contained 26 items. Factor analysis identified five themes of pacing contained within the APQ-26: Activity adjustment, Activity consistency, Activity planning, Activity acceptance and Activity progression.
  The APQ-26 has been modified for the purpose of this study with the addition of two items to correspond to important aspects of pacing that were not included in the APQ-26. The APQ-28 reflects the content of the activity pacing framework.
  The APQ-28 will be used to measure activity pacing at 3-months follow up after the end of the 6-week's programme.
  Each of the five themes of pacing is calculated as a mean score (0-4), where higher scores indicated more implementation of pacing strategies.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: Of the 107 participants who completed baseline data collection (T1) and those who completed the end of treatment (T2) data collection, 52 participants completed the 3-month follow-up data collection (T3). There were two missing answers for APQ Activity adjustment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 52
score on a scale
  APQ-28 Activity adjustment: number analyzed (Participants) | 50
  APQ-28 Activity adjustment | 2.33 (0.90)
  APQ-28 Activity planning | 2.06 (1.02)
  APQ-28 Activity consistency | 2.37 (0.72)
  APQ-28 Activity acceptance | 2.42 (0.95)
  APQ-28 Activity progression | 2.00 (0.91)

5. Secondary Outcome: Pain at Baseline: 11-point Numerical Rating Scale (NRS) of Pain
Description: Two 11-point Numerical Rating Scales (NRS) will assess current pain and usual pain, where 0='no pain' and 10='worst possible pain' at baseline (pre-treatment: up to one week before the programme)
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: 107 participants completed the baseline questionnaire booklet. However, there was one missing answer for Current pain (n=106); and four missing answers for Usual pain (n=103).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 106
score on a scale
  Current pain | 6.71 (1.96)
  Usual pain: number analyzed (Participants) | 103
  Usual pain | 7.47 (1.69)

6. Secondary Outcome: Pain at the End of Treatment (6-weeks): 11-point Numerical Rating Scale (NRS) of Pain
Description: Two 11-point Numerical Rating Scales (NRS) will assess current pain and usual pain, where 0='no pain' and 10='worst possible pain' at the end of the 6-week's programme.
Time Frame: 6-weeks (end of the programme)
Population: All 65 participants completed the scales for current and usual pain in the 6-weeks (T2) questionnaire booklet. There were no missing answers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 65
score on a scale
  Current pain | 5.31 (2.38)
  Usual pain | 6.62 (2.08)

7. Secondary Outcome: Pain at 3-months Follow up: 11-point Numerical Rating Scale (NRS) of Pain
Description: Two 11-point Numerical Rating Scales (NRS) will assess current pain and usual pain, where 0='no pain' and 10='worst possible pain' at 3-months follow up after the end of the 6-week's programme
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: 52 participants completed the questionnaire booklets at 3-months follow-up. However, there were two missing answers for Usual pain.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 52
score on a scale
  Current pain | 5.65 (2.31)
  Usual pain: number analyzed (Participants) | 50
  Usual pain | 6.54 (1.93)

8. Secondary Outcome: Depression at Baseline: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) contains nine items that screen for and measure the severity of depression in the clinical setting. Items are developed based on the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV). This will be measured at baseline (pre-treatment: up to one week before the programme). The total range of scores is 0-27, where 1-4=minimal depression, 5-9=mild depression, 10-14=moderate depression and ≥15=severe depression.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: Three missing answers from the 107 participants at baseline (T1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 104
score on a scale | 13.26 (6.86)

9. Secondary Outcome: Depression at the End of Treatment (6-weeks): Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) contains nine items that screen for and measure the severity of depression in the clinical setting. Items are developed based on the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV). This will be measured at the end of the 6-week's programme. The total range of scores is 0-27, where 1-4=minimal depression, 5-9=mild depression, 10-14=moderate depression and ≥15=severe depression.
Time Frame: 6-weeks (end of the programme)
Population: Two missing answers from the 65 participants at T2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 63
score on a scale | 7.14 (6.09)

10. Secondary Outcome: Depression at 3-months Follow-up: Patient Health Questionnaire-9
Description: The Patient Health Questionnaire (PHQ-9) contains nine items that screen for and measure the severity of depression in the clinical setting. Items are developed based on the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV). This will be measured at 3-months follow up after the end of the 6-week's programme. The total range of scores is 0-27, where 1-4=minimal depression, 5-9=mild depression, 10-14=moderate depression and ≥15=severe depression.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: One missing answer from the 52 participants at T3.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 51
score on a scale | 9.09 (5.76)

11. Secondary Outcome: Anxiety at Baseline: Generalised Anxiety Disorder Assessment (GAD-7)
Description: The Generalised Anxiety Disorder Assessment (GAD-7) contains seven items that screen for and measure the severity of anxiety in the clinical setting. The items are based on the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV). This will be measured at baseline (pre-treatment: up to one week before the programme). The total range of scores is 0-21, where 5-9=mild anxiety, 10-14=moderate anxiety and ≥15=severe anxiety.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: One missing answer from the 107 participants at baseline (T1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 106
score on a scale | 9.89 (5.92)

12. Secondary Outcome: Anxiety at the End of Treatment (6-weeks): Generalised Anxiety Disorder Assessment (GAD-7)
Description: The Generalised Anxiety Disorder Assessment (GAD-7) contains seven items that screen for and measure the severity of anxiety in the clinical setting. The items are based on the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV). This will be measured at the end of the 6-week's programme. The total range of scores is 0-21, where 5-9=mild anxiety, 10-14=moderate anxiety and ≥15=severe anxiety.
Time Frame: 6-weeks (end of the programme)
Population: 65 participants at 6-weeks data collection (T2)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 65
score on a scale | 5.40 (5.12)

13. Secondary Outcome: Anxiety at 3-months Follow up: Generalised Anxiety Disorder Assessment (GAD-7)
Description: The Generalised Anxiety Disorder Assessment (GAD-7) contains seven items that screen for and measure the severity of anxiety in the clinical setting. The items are based on the Diagnostic and Statistical Manual of Mental Disorders 4th Edition (DSM-IV). This will be measured at 3-months follow up after the end of the 6-week's programme. The total range of scores is 0-21, where 5-9=mild anxiety, 10-14=moderate anxiety and ≥15=severe anxiety.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: 52 participants provided data at 3-months (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 52
score on a scale | 6.10 (5.23)

14. Secondary Outcome: Self-efficacy at Baseline: Pain Self Efficacy Questionnaire (PSEQ)
Description: The Pain Self-Efficacy Questionnaire (PSEQ) contains 10 items that assess a persons' confidence in their ability to do things despite their pain. This will be measured at baseline (pre-treatment: up to one week before the programme). The range of total scores is 0-60 where PSEQ≥40 indicate those patients who are more likely to continue implementing coping strategies and PSEQ≤16 are considered low.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: All 107 participants at T1 provided an answer
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 107
score on a scale | 25.67 (11.93)

15. Secondary Outcome: Self-efficacy at the End of Treatment: Pain Self Efficacy Questionnaire (PSEQ)
Description: The Pain Self-Efficacy Questionnaire (PSEQ) contains 10 items that assess a persons' confidence in their ability to do things despite their pain. This will be measured at the end of the 6-week's programme. The range of total scores is 0-60 where PSEQ≥40 indicate those patients who are more likely to continue implementing coping strategies and PSEQ≤16 are considered low.
Time Frame: 6-weeks (end of the programme)
Population: All 65 participants at T2 provided an answer
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 65
score on a scale | 36.29 (14.12)

16. Secondary Outcome: Self-efficacy at 3-months Follow up: Pain Self Efficacy Questionnaire (PSEQ)
Description: The Pain Self-Efficacy Questionnaire (PSEQ) contains 10 items that assess a persons' confidence in their ability to do things despite their pain. This will be measured at 3-months follow up after the end of the 6-week's programme. The range of total scores is 0-60 where PSEQ≥40 indicate those patients who are more likely to continue implementing coping strategies and PSEQ≤16 are considered low.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: All 52 participants at 3-months follow-up (T3) provided an answer
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 52
score on a scale | 34.68 (14.26)

17. Secondary Outcome: Fatigue at Baseline: Chalder Fatigue Questionnaire (CFQ)
Description: The Chalder Fatigue Questionnaire (CFQ) contains two subscales: physical fatigue (seven items) and mental fatigue (four items). This will be measured at baseline (pre-treatment: up to one week before the programme). The total range for physical fatigue is 7-28 and the range for mental fatigue is 4-16, where higher scores indicated less fatigue.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: 107 participants completed the first questionnaire booklet (T1). However, there were four missing answers for physical fatigue (n=103) and one missing answer for mental fatigue (n-106)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 106
score on a scale
  Physical fatigue: number analyzed (Participants) | 103
  Physical fatigue | 14.81 (4.54)
  Mental fatigue | 8.83 (2.94)

18. Secondary Outcome: Fatigue at the End of Treatment: Chalder Fatigue Questionnaire (CFQ)
Description: The Chalder Fatigue Questionnaire (CFQ) contains two subscales: physical fatigue (seven items) and mental fatigue (four items). This will be measured at the end of the 6-week's programme. The total range for physical fatigue is 7-28 and the range for mental fatigue is 4-16, where higher scores indicated less fatigue.
Time Frame: 6-weeks (end of the programme)
Population: 65 participants completed the 6-weeks questionnaire booklet (T2). However, there were three missing answers on the Physical fatigue subscale (n=62) and one missing answer on the Mental fatigue scale (n=64).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 64
score on a scale
  Physical fatigue: number analyzed (Participants) | 62
  Physical fatigue | 20.31 (3.92)
  Mental fatigue | 11.28 (2.43)

19. Secondary Outcome: Fatigue at 3-months Follow up: Chalder Fatigue Questionnaire (CFQ)
Description: The Chalder Fatigue Questionnaire (CFQ) contains two subscales: physical fatigue (seven items) and mental fatigue (four items). This will be measured at 3-months follow up after the end of the 6-week's programme. The total range for physical fatigue is 7-28 and the range for mental fatigue is 4-16, where higher scores indicated less fatigue.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: Three missing answers for the Physical fatigue subscale; one missing answer for the Mental fatigue subscale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 51
score on a scale
  Physical fatigue: number analyzed (Participants) | 49
  Physical fatigue | 18.18 (4.16)
  Mental fatigue | 10.92 (2.34)

20. Secondary Outcome: Pain-related Anxiety, Fear and Avoidance at Baseline: Pain Anxiety Symptoms Scale-short Version (PASS-20)
Description: The Pain Anxiety Symptoms Scale-short version (PASS-20) measures pain-related fear, anxiety and avoidance and it contains four subscales: cognitive anxiety, escape/avoidance, fearful thoughts and physiological anxiety. This will be measured at baseline (pre-treatment: up to one week before the programme). Only the Escape/avoidance subscale data were analysed to provide an measure of avoidance. The total score of this 5 item subscale ranges from 0-25 where higher scores indicated greater avoidance.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: One missing answer
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 106
score on a scale | 13.14 (5.98)

21. Secondary Outcome: Pain-related Anxiety, Fear and Avoidance at the End of Treatment: Pain Anxiety Symptoms Scale-short Version (PASS-20)
Description: The Pain Anxiety Symptoms Scale-short version (PASS-20) measures pain-related fear, anxiety and avoidance and it contains four subscales: cognitive anxiety, escape/avoidance, fearful thoughts and physiological anxiety. This will be measured at the end of the 6-week's programme. Only the Escape/avoidance subscale data were analysed to provide an measure of avoidance. The total score of this 5 item subscale ranges from 0-25 where higher scores indicated greater avoidance.
Time Frame: 6-weeks (end of the programme)
Population: One missing answer
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 64
score on a scale | 10.28 (5.89)

22. Secondary Outcome: Pain-related Anxiety, Fear and Avoidance at 3-months Follow up: Pain Anxiety Symptoms Scale-short Version (PASS-20)
Description: The Pain Anxiety Symptoms Scale-short version (PASS-20) measures pain-related fear, anxiety and avoidance and it contains four subscales: cognitive anxiety, escape/avoidance, fearful thoughts and physiological anxiety. This will be measured at 3-months follow up after the end of the 6-week's programme. Only the Escape/avoidance subscale data were analysed to provide an measure of avoidance. The total score of this 5 item subscale ranges from 0-25 where higher scores indicated greater avoidance.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: All 52 participants at 3-months follow-up (T3) provided an answer for this subscale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 52
score on a scale | 12.12 (5.79)

23. Secondary Outcome: Physical and Mental Function at Baseline: 12-Item Short-Form Health Survey (SF-12)
Description: The 12-Item Short-Form Health Survey (SF-12) is a generic health survey that assesses physical and mental function. This will be measured at baseline (pre-treatment: up to one week before the programme). The two subscale scores have a maximum score of 100, where higher scores indicated better function.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: Two missing answers for the physical and mental function subscales
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 105
score on a scale
  Physical function | 33.96 (8.82)
  Mental function | 40.00 (11.36)

24. Secondary Outcome: Physical and Mental Function at the End of Treatment: 12-Item Short-Form Health Survey (SF-12)
Description: The 12-Item Short-Form Health Survey (SF-12) is a generic health survey that assesses physical and mental function. This will be measured at the end of the 6-week's programme. The two subscale scores have a maximum score of 100, where higher scores indicated better function.
Time Frame: 6-weeks (end of the programme)
Population: Two missing answers on the Physical and Mental function subscales
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 63
score on a scale
  Physical function | 38.82 (9.06)
  Mental function | 45.83 (11.48)

25. Secondary Outcome: Physical and Mental Function at 3-months Follow up: 12-Item Short-Form Health Survey (SF-12)
Description: The 12-Item Short-Form Health Survey (SF-12) is a generic health survey that assesses physical and mental function. This will be measured at 3-months follow up after the end of the 6-week's programme. The two subscale scores have a maximum score of 100, where higher scores indicated better function.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: Five missing answers on the Physical and Mental function subscales
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 47
score on a scale
  Physical function | 36.55 (9.81)
  Mental function | 44.56 (10.60)

26. Secondary Outcome: General Health Status and Quality of Life at Baseline: EuroQol (EQ-5D-5L)
Description: The EuroQol (EQ-5D-5L) is a generic measure of health status that is widely used to assess both clinical and economic efficacy; and to compare health status across diseases. This will be measured at baseline (pre-treatment: up to one week before the programme). The EQ-5D-5L was calculated as an index score (0-1) where higher scores indicate better health-related quality of life.
Time Frame: Baseline (pre-treatment: up to one week before the programme)
Population: Seven missing answers from the 107 participants at baseline (T1).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 100
score on a scale | 0.42 (0.25)

27. Secondary Outcome: General Health Status and Quality of Life at the End of Treatment: EuroQol (EQ-5D-5L)
Description: The EuroQol (EQ-5D-5L) is a generic measure of health status that is widely used to assess both clinical and economic efficacy; and to compare health status across diseases. This will be measured at the end of the 6-week's programme. The EQ-5D-5L was calculated as an index score (0-1) where higher scores indicate better health-related quality of life.
Time Frame: 6-weeks (end of the programme)
Population: Six missing answers from the 65 participants at 6-weeks (T2) data collection
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 59
score on a scale | 0.56 (0.28)

28. Secondary Outcome: General Health Status and Quality of Life at 3-months Follow up: EuroQol (EQ-5D-5L)
Description: The EuroQol (EQ-5D-5L) is a generic measure of health status that is widely used to assess both clinical and economic efficacy; and to compare health status across diseases. This will be measured at 3-months follow up after the end of the 6-week's programme. The EQ-5D-5L was calculated as an index score (0-1) where higher scores indicate better health-related quality of life.
Time Frame: 3-months follow-up (after the end of the 6-week's programme)
Population: Seven missing answers from the 52 participants who responded to the 3-months follow-up (T3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Activity Pacing Framework
Number analyzed (Participants) | 45
score on a scale | 0.52 (0.29)

ADVERSE EVENTS:
Time Frame: There were no adverse events throughout the duration of the study, that is, between the start of recruitment in May 2018 and the end of the 3-months follow-up data collection in December 2019.
Description: There were zero adverse events among a possible sample of 107 patients who commenced the rehabilitation programme; nor were there any adverse events during the interviews with the five healthcare professionals.
Arm/Group | Activity Pacing Framework
All-Cause Mortality (participants affected / at risk) | 0/107
Serious Adverse Events (participants affected / at risk) | 0/107
Other Adverse Events (participants affected / at risk) | 0/107

LIMITATIONS AND CAVEATS:
The target sample size of n=50 patients at 3-months follow-up (T3) for the feasibility study was attained (actual sample at T3: n=52). Despite recruiting to target for the feasibility study, this sample was not powered with a control arm to determine treatment effectiveness.

The generalisability of this study is limited to a sample of predominantly females, of white ethnic origin and recruited from only one Pain Service in Northern England, United Kingdom (UK).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT03497585/Prot_SAP_002.pdf
  • Informed Consent Form (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT03497585/ICF_003.pdf